CLINICAL TRIAL: NCT06431854
Title: The Efficacy, Efficiency, and Patient Experience of a New Intensive Treatment Program for Adolescents With High-complexity Eating Disorders: MINERVA
Brief Title: Evaluation of a New Treatment Program for Adolescents With Eating Disorders: MINERVA Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: University Ramon Llull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MINERVA
Record Dates: First submitted 2024-04-12; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Eating Disorders in Adolescence; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Other Specified Feeding or Eating Disorder
Keywords: Eating Disorders; Adolescence; Inpatient treatment; Home treatment; Cognitive Behaviorial Therapy; Family-Based Treatment; Dialectical Behavioral Therapy; Systemic Family Treatment
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: This study will compare prospective data with retrospective data of patients that followed Treatment As Usual (TAU). Treatment As Usual (TAU) involves arranging visits for external consultations, partial hospitalization, and inpatient admissions as necessary, by following clinical guidelines. The retrospective control group consists of 60 patients, matched in age, sex, Body Mass Index (BMI), and diagnosis of eating disorder (ED) with the prospective group. Subjects are identified by reviewing medical records of patients treated at the ED unit of Hospital Sant Joan de Déu before the initiation of the MINERVA program. The temporal reference is the first day of admission to acute total hospitalization. Subjects present the same criteria of poor treatment response as the prospective group, ensuring severity comparability with the prospective group. Exclusion occurs if there is ≥20% missing data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient group (Experimental): This group comprises 60 patients aged 12 to 17 diagnosed with an eating disorder. They must have shown poor response to treatment, defined as having one of the two conditions: 1) undergoing over a year of treatment, including partial and total hospitalization, without symptom stabilization (needing high-intensive treatment units i.e. not being able to follow individual treatment in external consultations); 2) having more than three admissions without symptom stabilization in less than one year. They will be recruited from child/adolescent ED units in Catalonia. Exclusions will be acute ED pathology requiring urgent pediatric attention or admission to an acute psychiatric ward.
  Interventions: Behavioral: ED-MINERVA Program

INTERVENTIONS:
Behavioral: ED-MINERVA Program — ED-MINERVA Program aims to improve ED symptoms and related difficulties of the patient and provide tools to enhance the family's management (nutritionally, emotionally, and behaviorally) in their natural environment. The treatment consists of four phases with a gradually decreasing therapeutic intensity, ranging from total hospitalization, family treatment apartment, to home treatment and subsequent linkage with specialized local facilities. The ED-MINERVA program uses various aspects of family-based treatment, cognitive behavioral therapy, dialectical behavioral therapy, and systemic family therapy.

SUMMARY:
The aim of this study is to investigate the efficacy, efficiency, and patient experience of a new intervention program on adolescents with high-complexity eating disorders (ED). A prospective group of adolescents with ED (N=60) will follow this treatment program including four different phases: 1) Inpatient treatment; 2) Family Treatment Apartment; 3) Home Treatment; 4) Recovery within the community. The investigators will use a retrospective, control group (N=60) that matched the prospective group in age, sex, ED diagnosis, and severe symptomatology. Primary variables regarding Body Mass Index (BMI), ED symptomatology, functionality, recovery (yes/no), type of outpatient services (low/mid/high intensity), number of readmissions, and patient experience will be assessed at discharge, and after 6 and 12 months. Secondary variables include anxiety, depression, readiness to recover, quality of life symptoms, caregiver skills, and functionality of the family

DETAILED DESCRIPTION:
The goal of this single-center, longitudinal study is to test the efficacy, efficiency, and patient experience of a new intensive treatment program in adolescents with high-complex eating disorders. The main questions it aims to answer are:

* What are the efficacy, efficiency, and patient experiences (families and patients) of the new treatment program in adolescents with high-complex eating disorders?
* What are the long-term effects of efficacy and efficiency (after 6 and after 12 months) of the new treatment program in adolescents with high-complex eating disorders?

Participants will receive this new treatment program in four different phases between 16 and 20 weeks approximately.

* 1st: inpatient treatment (4 weeks): Set-up: inpatient ED unit at the hospital (without the family). Objectives: maintenance of physical stabilization; ensuring adequate food intake while preventing compensatory behaviors; addressing ED-related problems; improving nutritional administration; enhancing awareness of the disorder and motivating the patient to change.
* 2nd: family treatment apartment (2-3 weeks): Set-up: apartments where patients and their families live together that is owned by the healthcare system provider. Family treatment apartments are within a hospital context to facilitate a good transition to home treatment.

Objectives: intensifying the treatment within a hospital setting that targets the difficulties the family encounter in managing ED symptoms; intervening from a systemic perspective; involving other family members in the treatment; collaborating with the family in developing skills to cope with the disorder; working on more autonomy and improved ED decision-making; facilitating the transition from hospitalization to home; facilitate access to the hospital staff and leads to a high frequency treatment.

* 3rd: home treatment (8-9 weeks): Set-up: Patients live in their own home. Objectives: facilitating a good transition from hospitalization and family treatment apartments to home; generalize psychological skills and learnings; assisting in the progress that began in the hospital environment; providing treatment in a more family and social context; empowering families in their natural setting; promoting integration of the patient into their family, social, and school environments.
* 4th: Recovery within the community (2-4 weeks): Set-up: transferring to the patients' specialized ED reference center. Objectives: gradually reducing the intervention from MINERVA; promoting autonomy and emotional management within their family and school environment; ensuring continued care with their ED reference unit; monitoring the implemented intervention.

The current model will provide different treatment models during these phases.

* family-based treatment
* cognitive behavioural therapy
* dialectical behavioural therapy
* systemic family therapy

ELIGIBILITY:
Inclusion Criteria for the prospective experimental group:

* Patient diagnosed with an Eating Disorder (according to the DSM-5) through a semi-structured interview (K-SADS PL-5)
* Aged between 12 and 17 years old
* Both patients and parents are willing to participate in the study and sign the informed consent to accept participation
* Patient with a poor response to treatment, defined as having one of the following two conditions:

  1. undergoing over a year of treatment, including partial and total hospitalization, without symptom stabilization, experiencing severe psychological distress, eating symptomatology, comorbidities, or family dysfunction during this period (clinical improvement of at least 50 on the CGAS functioning scale) OR
  2. undergoing more than three admissions without symptom stabilization (clinical improvement of at least 50 on the CGAS functioning scale).

     Exclusion criteria for the prospective group:
* Acute ED pathology and biological decompensation that require urgent pediatric attention or admission to an acute psychiatric ward.

Inclusion criteria for the retrospective control group:

* Aged between 12 and 17 years old
* Diagnosed with an Eating Disorder (according to the DSM-5)
* Received treatment in Sant Joan de Déu between 2012 and 2022
* Patient with a poor response to treatment, defined as having one of the following two conditions:

  1. undergoing over a year of treatment, including partial or total hospitalization, without achieving stabilization of ED symptomatology (needing high-intensive treatment units i.e. not being able to follow individual treatment in external consultations) OR
  2. undergoing more than three admissions without symptom stabilization once referred to partial hospitalization in less than one year, including a similar psychological state and characteristics as the first condition

Exclusion criteria for the retrospective control group:

* Missingness of 20% or more of the required data

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
O1: Changes in BMI (efficacy) | Up to 20 weeks
  Evaluate the change in BMI between the beginning and the end of the intervention of the patients included in the MINERVA program. Furthermore, BMI changes of the MINERVA group will be compared with retrospective data. Weight in kilograms and height in meters will be combined to report BMI in kg/m^2. Improvements in O1 and O2 need to be detected to consider the MINERVA program effective. Additionally, improvements in at least one of the other two outcomes (O3 and/or O4) need to be detected to conclude that the MINERVA program is effective at clinical and functional levels, in comparison to previous treatment programs.
O2: Changes in clinical eating symptomatology (efficacy) | Up to 20 weeks
  Evaluate the changes in clinical eating symptomatology between the beginning and the end of the intervention of patients included in the MINERVA program. The Eating Disorder Inventory 3 (EDI-3) will be used to assess clinical eating symptomatology. It comprises 91 items where responses are given on a Likert scale (0-4). The subscales regarding 'drive for thinness' and 'body dissatisfaction' will be used for the main objective, where improvements in both subscales need to be detected. Improvements in O1 and O2 need to be detected to consider the MINERVA program effective. Additionally, improvements in at least one of the other two outcomes (O3 and/or O4) need to be detected to conclude that the MINERVA program is effective at clinical and functional levels, in comparison to previous treatment programs.
O3: Changes in functionality of the patient (efficacy) | Up to 20 weeks
  Evaluate the functionality of the patient between the beginning and the end of the intervention in patients included in the MINERVA program. Functionally will also be assessed at 6 and 12 months after completing the program. The Children's Global Assessment Scale (CGAS) will be used to assess functionality. CGAS is scored on a range from 1 to 100, whereby a higher score indicates a better outcome. Improvements in O1 and O2 need to be detected to consider the MINERVA program effective. Additionally, improvements in at least one of the other two outcomes (O3 and/or O4) need to be detected to conclude that the MINERVA program is effective at clinical and functional levels, in comparison to previous treatment programs.
O4: Changes in recovery rates (efficacy) | 6 months after treatment completion
  Evaluate the percentage of patients who do no longer meet diagnostics criteria for a primary eating disorder. Furthermore, data will be compared with retrospective data. Improvements in O1 and O2 need to be detected to consider the MINERVA program effective. Additionally, improvements in at least one of the other two outcomes (O3 and/or O4) need to be detected to conclude that the MINERVA program is effective at clinical and functional levels, in comparison to previous treatment programs.
O5: Percentage of patients in low-intensity care settings (efficiency) | 6 months after treatment completion
  Determine the percentage of patients in low-intensity care settings after 6 months of completing the program (including day hospital and specific outpatient consultations). The MINERVA program will be considered efficient if more than 60% of the patients will be able to continue treatment at low-intensity outpatient services (including day hospitals and specific external consultations) in ED units or community resources.
Percentages of readmissions (efficiency) | 6 months after treatment completion
  Determine the percentage of readmissions at 6 and 12 months after completing the program. Furthermore, this data will be compared with retrospective data. The MINERVA program will be considered efficient if more than 60% of the patients will be able to continue treatment at low-intensity outpatient services (including day hospitals and specific external consultations) in ED units. Furthermore, the program will be considered more efficient than TAU if significant lower readmission percentages in O6 and O7 will be detected.
Percentages of readmissions (efficiency) | 12 months after treatment completion
  Determine the percentage of readmissions at 6 and 12 months after completing the program. Furthermore, this data will be compared with retrospective data. The MINERVA program will be considered efficient if more than 60% of the patients will be able to continue treatment at low-intensity outpatient services (including day hospitals and specific external consultations) in ED units. Furthermore, the program will be considered more efficient than TAU if significant lower readmission percentages in O6 and O7 will be detected.
Patient experience | Up to 20 weeks
  Evaluate the level of satisfaction with the received intervention, adherence, and the rate of patient and family dropout (less than 20%). Patient Experience will be assessed through individual interviews with the patient and their family, and Patient-Reported Experience Measures (PREMs) surveys. PREM is a systematic online survey that assesses and describes the experience regarding healthcare services. The survey consists of Likert-scale and open-ended questions to gather narrative information that enriches qualitative data with more details and context.

SECONDARY OUTCOMES:
Changes in symptoms of anxiety | Up to 20 weeks
  Evaluate changes in symptoms of anxiety between the beginning and the end of the intervention of the patients included in the MINERVA program. The State-Trait Anxiety Inventory (STAI) will be used to assess anxiety. STAI is scored on a range from 20 to 80, whereby a higher score indicates a worse outcome.
Changes in symptoms of depression | Up to 20 weeks
  Evaluate changes in symptoms of depression between the beginning and the end of the intervention of the patients included in the MINERVA program. The Beck Depression Inventory (BDI) will be used to assess depression. It consists of 21 Likert-scale items, ranging from 0 to 3, with a cutoff point of 13 or higher that indicates the presence of depressive symptoms.
Changes in readiness to recover | Up to 20 weeks
  Evaluate changes in readiness to recover between the beginning and the end of the intervention of the patients included in the MINERVA program. The Anorexia Nervosa Stages of Change Questionnaire (ANSOCQ) will be used to assess motivation of recovering. It consist of 20 Likert-scale items, ranging from 1 to 5, whereby a higher score indicates a better outcome.
Changes in caregiver skills | Up to 20 weeks
  Assess caregiver skill changes in the families of the included patients. The Caregiver Skills (CASK) will be used to assess caregiver skills. CASK is scored on a range from 0 to 100, whereby a higher outcome indicates a better outcome.
Changes in quality of life | Up to 20 weeks
  Examine changes in the quality of life of the patients and their families. The Kidscreen-27: Quality of Life Inventory will be used to assess the quality of life. It consists of 27 Likert-scale items, ranging from 1 to 5, whereby a higher score indicates a better outcome.
Functionality of the patient | 6 months after treatment completion
  Evaluate the functionality of the patient between the beginning and the end of the intervention in patients included in the MINERVA program. Functionally will also be assessed at 6 and 12 months after completing the program. The Children's Global Assessment Scale (CGAS) will be used to assess functionality. CGAS is scored on a range from 1 to 100, whereby a higher score indicates a better outcome.
Functionality of the patient | 12 months after treatment completion
  Evaluate the functionality of the patient between the beginning and the end of the intervention in patients included in the MINERVA program. Functionally will also be assessed at 6 and 12 months after completing the program. The Children's Global Assessment Scale (CGAS) will be used to assess functionality. CGAS is scored on a range from 1 to 100, whereby a higher score indicates a better outcome.
Mental illness in parents | Up to 20 weeks
  Mental illness in parents will be assessed at the beginning and the end of the intervention. The Kiddie Schedule For Affective Disorders and Schizophrenia-Present and Lifetime 5 (K-SADS-PL-5) will be used to assess mental illness in parents. The K-SADS-PL-5 is a semi-structured diagnostic interview designed to clinically diagnose ED and identify psychiatric comorbidities. It includes an introductory interview, a screening interview, and diagnostic supplements.
Parental skills in managing eating disorders | Up to 20 weeks
  Skills in managing eating disorders of the parents will be assessed at the beginning and the end of the intervention. The Caregiver Skills (CASK) will be used to assess caregiver skills. CASK is scored on a range from 0 to 100, whereby a higher score indicates a better outcome.
Functionality and dynamics of the family | Up to 20 weeks
  The functionality and dynamics of the family will be assessed at the beginning and the end of the intervention. The SCORE-15 will be used to assess changes in functionality and dynamics. SCORE-15 is a self-administered questionnaire that consists of 15 Likert-type items (1-5) and is divided into three scales: strengths and adaptability, concerns or distress, and communication difficulties. The total score can be on a range from 15 to 75, whereby a higher score indicates a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Serrano-Troncoso, Dr., Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through the current study may be provided to qualified researchers with academic interest in eating disorders. Data shared will be encoded, with no Protected Health Information (PHI) included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted immediately following publication. There will be no end date.
Access Criteria: Proposals should be directed to the Principal Investigator. To obtain access, data requestors will need to sign a data agreement with our institution, to comply with legal requirements and data protection rights. The study protocol and/or amendment to the protocol will be reviewed by the corresponding Ethics Committees.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT06431854/Prot_SAP_000.pdf